CLINICAL TRIAL: NCT00401752
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Parallel-group, 8 Week Comparative Efficacy and Safety Study of Esomeprazole 20 mg Every Day (qd) Versus Ranitidine 150 mg Twice a Day (Bid) in Patients With an NSAID-associated Gastric Ulcer When Daily NSAID is Continued
Brief Title: Efficacy and Safety Study of Esomeprazole 20mg qd vs Ranitidine 150mg Bid in Patients With an NSAID-induced Gastric Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9617L00001
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-06

CONDITIONS: Gastric Ulcer
Keywords: NSAID-associated gastric ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — Esomeprazole; Ranitidine

INTERVENTIONS:
Drug: Esomeprazole
Drug: Ranitidine

SUMMARY:
The purpose of this study is to assess the efficacy of esomeprazole 20 mg dosed once daily and ranitidine 150 mg dosed twice daily through 4 weeks of treatment for the healing of gastric ulcers in patients receiving daily non-steroidal anti-inflammatory drug (NSAID)therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* A clinical diagnosis of a chronic condition that requires daily NSAID treatment for at least 2 months.
* Daily NSAID dose and type must have been stable for at least 2 weeks prior to the baseline endoscopy;orally;

Exclusion Criteria:

* History of esophageal, gastric or duodenal surgery, except for simple closure of an ulcer.
* History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2006-03; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca
Locations (9):
- China (8):
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Suzhou, Jiangsu
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi’an, Shanxi
  - Research Site, Beijing
  - Research Site, Shanghai
- Research Site, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 219 patients from 18 centers in China who had been receiving a stable daily dose of 1 or more NSAIDs for at least 2 weeks and who had an NSAID-associated GU verified by EGD at baseline were randomized. The first patient was enrolled on 31 Mar 2006, the last patient was completed on 17 Nov 2008.
Pre-assignment Details: Total 397 patients from 24 centers in China were enrolled. 178 patients were not randomised due to unwillingness to continue the study or development of any exclusion criteria, etc. Total 219 patients were randomised, 217 patients were included in ITT population.
Groups:
- Esomeprazole: Esomeprazole 20 mg tablet qd oral administration
- Ranitidine: ranitidine 150 mg capsule bid oral administration
Period: Overall Study
Arm/Group | Esomeprazole | Ranitidine
Started | 107 | 112
Number of Patients Received Treatment | 107 | 111
Patients Included in ITT Population | 106 | 111
Patients Included in Safety Population | 107 | 110
Patients Included in Per-Protocol Popula | 100 | 99
Completed | 97 | 94
Not Completed | 10 | 18
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Development of any exclusion criteria | 4 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Ranitidine | Total
Number analyzed (Participants) | 106 | 111 | 217
Age Continuous [Mean (Standard Deviation); unit: year] | 49.7 (11.01) | 50.9 (10.2) | 50.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 55 | 58 | 113

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Whose Gastric Ulcer(s) (GUs) Was (Were) Healed at Week 4 After Treatment With Esomeprazole 20 mg qd and Ranitidine 150 mg Bid in Patients Receiving Daily Non-steroidal Anti-inflammatory Drug (NSAID)Therapy.
Description: Healed was defined as the absence of gastric ulcers. It was calculated as the proportion of subjects whose gastric ulcer(s) healed after 4 weeks treatment.
  (Ulcers were on S stage, stage 1 = Nonblanchable erythema of intact skin, stage 2 = Partial thickness skin loss involving epidermis, dermis, or both, stage 3 = Full thickness skin loss involving damage to or necrosis of subcutaneous tissue, stage 4 = Full thickness skin loss with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures or absent).
Time Frame: 4 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 106 | 111
Percentage of participants | 59.4 | 59.5

2. Secondary Outcome: The Percentage of Subjects Whose Gastric Ulcer(s) Was (Were) Healed at Week 8 After Treatment With Esomeprazole 20 mg qd and Ranitidine 150 mg Bid in Patients Receiving Daily NSAID Therapy.
Description: Healed was defined as the absence of gastric ulcers (Ulcers were on S stage or absent). It was calculated as the proportion of subjects whose gastric ulcer(s) healed after 8 weeks treatment.
Time Frame: 8 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 106 | 111
Percentage of participants | 81.1 | 73.9

3. Secondary Outcome: The Resolution of Heartburn Symptoms at Week 4 and Week 8 After Treatment With Esomeprazole 20 mg qd and Ranitidine 150 mg Bid in Patients Receiving Daily NSAID Therapy.
Description: Resolution rate of investigator-assessed GI symptoms, including heartburn, acid regurgitation, nausea, abdominal fullness and sleep disorder. It was calculated as the percentage of subjects whose heartburn symptoms were resolved at Week 8.
Time Frame: week 4 and week 8
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 106 | 111
Percentage of participants | 100 | 97.7

4. Secondary Outcome: Percentage of Participants With the Occurance of Any Adverse Event.
Description: Safety evaluation including vital signs, physical examination, ECG, adverse events and clinical laboratory evaluations during 8 weeks treatment.
Time Frame: 8 weeks
Population: Patients included in safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 107 | 110
Percentage of participants | 16.8 | 22.7

5. Secondary Outcome: The Percentage of Participants Whose Duodenal Ulcer(s) (DUs) Was (Were) Healed at Week 4 and Week 8 After Treatment With Esomeprazole 20 mg qd and Ranitidine 150 mg Bid in Patients Receiving Daily NSAID Therapy.
Description: Healed was defined as the absence of ulcers (Ulcers were on S stage or absent). It was calculated as the proportion of subjects whose duodenal ulcer healed after 4 and 8 weeks treatment.
Time Frame: 4 and 8 week
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 15 | 22
Percentage of participants | 93.3 | 81.8

6. Secondary Outcome: The Percentage of Participants Whose GU(s) and DU(s) in Combination Were Healed at Week 4 and Week 8 After Treatment With Esomeprazole 20 mg qd and Ranitidine 150 mg Bid in Patients Receiving Daily NSAID Therapy
Description: Healed was defined as the absence of ulcers (Ulcers were on S stage or absent). It was calculated as the proportion of subjects whose gastric and duodenal ulcer healed after 4 and 8 weeks treatment.
Time Frame: 4 & 8 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole | Ranitidine
Number analyzed (Participants) | 106 | 111
Percentage of participants | 80.2 | 69.4

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Ranitidine
Serious Adverse Events (participants affected / at risk) | 2/107 | 2/110
Other Adverse Events (participants affected / at risk) | 13 | 16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=107) | Ranitidine (N=110)
Gastric Cancer (Gastrointestinal disorders) | 2 | 0
GU Haemorrhage (Gastrointestinal disorders) | 0 | 1
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Esomeprazole | Ranitidine
Dizziness (Nervous system disorders) | 0/107 | 5/110
Gastritis erosive (Gastrointestinal disorders) | 3/107 | 4/110
Alanine aminotransferase increased (Hepatobiliary disorders) | 2/107 | 0/110
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2/107 | 0/110
Gastric ulcer (Gastrointestinal disorders) | 2/107 | 1/110
Abdominal pain upper (Gastrointestinal disorders) | 1/107 | 2/110
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1/107 | 2/110
Duodenal ulcer (Gastrointestinal disorders) | 0/107 | 2/110
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/107 | 0/110

LIMITATIONS AND CAVEATS:
According to the protocol, the sample size was 320 patients which could achieve 80% power of superiority. Since the patient recruitment is very difficult, total 219 patients were randomized in present study, the power decreased to 60%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less